CLINICAL TRIAL: NCT01061034
Title: The Effect of Proton Pump Inhibitor (Omeprazole) on Acetosalisylic Acid Absorption.
Brief Title: Pharmacological Study That Measures Omeprazole Effect on Aspirins Absorption in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: dr. keren doenyas barak, internal medicine A asaf-harofeh medical center
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 180/07
Record Dates: First submitted 2009-05-03; First posted 2010-02-02 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2009-11

CONDITIONS: Aspirin Blood Level; Proton Pump Inhiditor Treatment
Keywords: pharmacokinetics; aspirin; proton pump inhiditor
MeSH Terms: interventions — Aspirin; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: aspirin and omeprazole — aspirin 100 mg, once daily aspirin 100 mg and omeprazole 20 mg both once daily.

SUMMARY:
Aspirin is a weak acid that crosses the gastric and intestinal mucosa by passive diffusion while in its lipophilic nature.Omeprazole, a proton pump inhibitor, inhibits gastric acid secretion.

We assumed that omeprazole inhibits aspirin absorption, thus reducing its action on platelets.

healthy volunteers, with no known peptic disease or bleeding disorders will be enrolled.

All volunteers will receive 7 days of Aspirin (100mg) alone, followed by 14 days of Aspirin and Omeprazole 20mg twice daily for 3 days and then 20mg once daily.

Blood levels of Aspirin will be determined by High performance liquid chromatography (HPLC), 0, 1, 2, 4, 6, 10, 24 hours after the administration of Aspirin alone on day 7 and Aspirin plus Omeprazole on day 21.

Platelet function tests will be determined by platelet-rich plasma aggregometry in response to Arachidonic acid (500mg/ml), Ristocetin (1.5mg/ml) and Adenosine 5'-diphosphate (20mM) on day 0 as baseline and on day 7 and 21 of the study.

ELIGIBILITY:
Inclusion Criteria:

-healthy volunteers

Exclusion Criteria:

* pretreatment with aspirin
* pretreatment with non steroidal anti inflamatory drugs
* pretreatment with antacids
* history of peptic ulcer disease
* coagulation or aggregation disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ahuva golik, prop., Study Director — asaf-harofemedical center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel

RESULTS

PARTICIPANT FLOW:
Recruitment Details: healthy volunteers were recruted on march 2007. all of the patients are co-workers in the department of medicine in assaf harofeh medical center.
Pre-assignment Details: one volunteer was excluded before enrollment due to recent consumption of NSAIDS
Groups:
- Aspirin Then Aspirin Plus Omeprazole: 7 days of Aspirin (100mg) alone, followed by 14 days of Aspirin and Omeprazole (20mg BID for 3 days and then 20mg once daily
Period: Aspirin
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Started | 9
Completed | 9
Not Completed | 0
Period: Aspirin Plus Omeprazole
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Aspirin Level in Blood (Area Under the Curve)
Description: Aspirins pharmacokinetics: aspirin blood level determined by use of high performance liquid chromatography (HPLC) at baseline, 1, 2,4,6,10 and 24 hours after administration of aspirin on day 7 and on day 21.
  The area unther the time vs. concentration curve of the reccurent measurments(AUC) reflects bioavailability of aspirin.
Time Frame: on day 7,on day 21
Population: 9 volunteers completed the study, one volunteer was excluded from pharmacokinetics, because serum salicylic acid concentration was not at the baseline (non-detectable) in the 0-hour sample.
Measure: Mean (Standard Deviation); unit: mg*hour/mL
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Number analyzed (Participants) | 8
mg*hour/mL
  aspirin area under the curve on day 7 | 49.4 (13.5)
  aspirin area under the curve on day 21 | 50.7 (15.3)
  1 hour after admission day 7 (aspirin alone) | 8.7 (4)
  1 hour after admission day 21 (aspirin+omeprazole) | 6.5 (4.1)

2. Secondary Outcome: Platelet Function Tests
Description: Platelet function tests were determined by optical whole blood aggregometry in response to arachidonic acid and adenosine diphosphate.
  the results reflects the percent of active platelets.
Time Frame: on day 0 as a baseline and on day 7 and 21 of the study.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Number analyzed (Participants) | 9
percent
  day 0 | 80 (4.18)
  day 7 | 8.55 (2.45)
  day 21 | 8.77 (2.38)

ADVERSE EVENTS:
Arm/Group | Aspirin Then Aspirin Plus Omeprazole
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 1/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aspirin Then Aspirin Plus Omeprazole (N=9)
mild dyspepsia (Gastrointestinal disorders) | 1 — one volunteer complained mild dyspepsia unther aspirin treatment alone. his complaine resolved withoud any special intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No